CLINICAL TRIAL: NCT04882813
Title: Replication of the DAPA-CKD (Chronic Kidney Disease) Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-DAPA-CKD
Record Dates: First submitted 2021-05-04; First posted 2021-05-12 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — dapagliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dapagliflozin: Exposure group
  Interventions: Drug: Dapagliflozin
- Sitagliptin: Reference group
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin dispensing claim is used as the exposure group.
  Groups: Dapagliflozin
Drug: Sitagliptin — Sitagliptin dispensing claim is used as the reference group.
  Groups: Sitagliptin

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates through standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Inclusion Criteria:

* 18 years of age [Day 0, Day 0]
* eGFR ≥25 and ≤75 mL/min/1.73 m2 (CKD-EPI formula) at visit 1 (- All Time, Day 0]
* Evidence of increased albuminuria for 3 months or more before visit 1 and UACR ≥200 and ≤5000 mg/g at visit 1(- All Time, Day 0]
* Stable, and for the patient maximum tolerated labelled daily dose, treatment with ACEi or ARB for at least 4 weeks before visit 1, if not medically contraindicated (-All Time, Day -45]

Exclusion Criteria:

* Type I diabetes mellitus (-All Time, Day 0]
* Autosomal dominant or autosomal recessive polycystic kidney disease, lupus nephritis or Antineutrophil cytoplasmic antibody (ANCA) - associated vasculitis (-All Time, Day 0]
* Receiving cytotoxic therapy, immunosuppressive therapy or other immunotherapy for primary or secondary renal disease within 6 months prior to enrollment [Day -180, Day 0]
* NYHA class IV congestive heart failure at the time of enrollment [Day -180, Day 0]
* MI, unstable angina, stroke, transient ischemic attack within 8 weeks prior to enrollment [ Day -56, Day 0]
* Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) or valvular repair/replacement within 8 weeks prior to enrollment [Day -56, Day 0]
* Any condition outside the renal and cardiovascular study area with a life expectancy of <2 years based on investigator's clinical judgement [Day 0, Day 0]
* Hepatic impairment [aspartate transaminase or alanine transaminase >3 times the upper limit of normal (ULN) or total bilirubin >2 times the ULN at the time of enrollment] (- All Time, Day 0]
* History of organ transplantation (- All Time, Day 0]
* Receiving therapy with SGLT2 inhibitor within 8 weeks prior to enrollment or previous intolerance of an SGLT2 inhibitor [Day -56, Day -1]
* Exclude patients that have AKI, CKD V, ESRD and are on HD/PD during the baseline period [Day -14, Day 0] for AKI and [Day -180, Day 0] for CKD, ESRD, or Hemodialysis/Peritoneal Dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, retrospective cohort study design comparing dapagliflozin to sitagliptin. Although the trial compared dapagliflozin to placebo, for the current emulation we used an active comparator, sitagliptin, which is a dipeptidyl peptidase - (DPP-4) inhibitor. This is because both dapagliflozin and sitagliptin are guideline recommended as second to third line therapies used for the treatment of type 2 diabetes at the same stage of the disease and sitagliptin is not expected to have an effect on the primary outcome.
Sampling Method: Non-Probability Sample
Enrollment: 87727 (Actual)
Dates: Start 2020-12-13 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Relative hazard of the composite of end-stage renal disease or all-cause mortality | To study completion or censoring, up to 32 months
  Claims-based algorithm: see attached protocol for full definition

SECONDARY OUTCOMES:
Relative hazard of end-stage renal disease | To study completion or censoring event, up to 32 months
  Claims-based algorithm: see attached protocol for full definition
Relative hazard of all-cause mortality | To study completion or censoring event, up to 32 months
  Claims-based algorithm: see attached protocol for full definition

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT04882813/Prot_SAP_001.pdf